CLINICAL TRIAL: NCT06950658
Title: Breastfeeding Success in Term Newborn and Time of First Meconium Passage
Brief Title: Breastfeeding Success and Time of First Meconium Passage
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Other Study IDs: ATADEK 2023-16/554
Record Dates: First submitted 2025-04-21; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Meconium; Breastfeeding
Keywords: Breastfeeding; Breast milk; meconium passage; newborn; infant
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Term infants followed for breastfeeding success and time of first meconium passage: Data on the timing of first meconium passage to newborns were obtained and recorded by observing infants until discharge. Data on breastfeeding success in all their mother was assessed using the LATCH Breastfeeding Assessment Tool at three different time points: during the first breastfeeding session (0-1 hours), on day 1 (1-24 hours), and on day 2 (24-48 hours).

SUMMARY:
To investigate the relationship between breastfeeding success and the time of first meconium passage in term newborns.

DETAILED DESCRIPTION:
The timing of the first meconium passage in neonates is a useful indicator of distal colon function. Delayed passage may signal congenital distal bowel dysfunctions such as hirschsprung disease (HD), anorectal malformations, distal intestinal atresia, prematurity, or hypothyroidism. Several factors may influence the timing of the first meconium passage, including gestational age, birth weight, sex, mode of delivery, and presence of respiratory distress. Another significant factor is breastfeeding. Effective breastfeeding is known to contribute to the maturation of the gut microbiota and has long-term positive outcomes for both mother and infant. However, the literature lacks studies examining the relationship between breastfeeding and the timing of meconium passage.This study aimed to investigate the relationship between breastfeeding success and the timing of first meconium passage in term newborns. The following hypotheses were tested: (a) There is a relationship between breastfeeding success and the timing of meconium passage in term newborns; (b) Term newborns with higher breastfeeding success will pass meconium earlier.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term newborns (≥37 weeks gestation) who were exclusively breastfeed

Exclusion Criteria:

* Newborns who received any feeding other than direct breastfeeding (e.g., bottle, cup, etc.)

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consisted of all term newborns monitored in the postnatal period, while the sample comprised newborns who met the inclusion criteria and were followed in the Neonatal Care Unit.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Timing of the first meconium passage | The difference from the time of birth to the first observed meconium passage during hospitalization, assessed up to the time of discharge (up to 72 hours)
  Newborns were observed from birth until discharge. During this observation, when the first meconium passage occurred, the timing of meconium passage was recorded.
LATCH score | LATCH score assessed first breastfeeding, on day 1 (1-24 hours), and on day 2 (24-48 hours). The change in these time intervals will be assessed.
  Breastfeeding success in all newborns was assessed using the LATCH Breastfeeding Assessment Tool at three different time points: during the first breastfeeding session (0-1 hours), on day 1 (1-24 hours), and on day 2 (24-48 hours). The LATCH Breastfeeding Assessment Tool was developed in 1993 by Deborah Jensen and Sheila Wallace. The Turkish adaptation and validation of the tool were conducted by Yenal and Okumuş. Modeled after the Apgar scoring system, this tool was designed to objectively evaluate breastfeeding success, identify potential issues, and establish a standardized language among healthcare professionals. The scale consists of five criteria, each scored from 0 to 2, for a total score ranging from 0 to 10. Higher LATCH scores indicate greater breastfeeding success.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma IK, Byrne A. Early initiation of breastfeeding: a systematic literature review of factors and barriers in South Asia. Int Breastfeed J. 2016 Jun 18;11:17. doi: 10.1186/s13006-016-0076-7. eCollection 2016. PMID 27330542
- [Background] Feldman-Winter L, Kellams A, Peter-Wohl S, Taylor JS, Lee KG, Terrell MJ, Noble L, Maynor AR, Meek JY, Stuebe AM. Evidence-Based Updates on the First Week of Exclusive Breastfeeding Among Infants >/=35 Weeks. Pediatrics. 2020 Apr;145(4):e20183696. doi: 10.1542/peds.2018-3696. Epub 2020 Mar 11. PMID 32161111
- [Background] Ezomike UO, Ugwu EO, Ezomike NE, Eke CB, Ekenze SO. Evaluation of Impact of Perinatal Factors on Time to First Meconium Passage in Nigerian Neonates. Malawi Med J. 2019 Jun;31(2):150-154. doi: 10.4314/mmj.v31i2.8. PMID 31452849
- [Background] Bekkali N, Hamers SL, Schipperus MR, Reitsma JB, Valerio PG, Van Toledo L, Benninga MA. Duration of meconium passage in preterm and term infants. Arch Dis Child Fetal Neonatal Ed. 2008 Sep;93(5):F376-9. doi: 10.1136/adc.2008.138024. Epub 2008 Feb 19. PMID 18285377